CLINICAL TRIAL: NCT04249947
Title: A Phase 1 Dose Escalation and Expanded Cohort Study of P-PSMA-101 in Subjects With Metastatic Castration-Resistant Prostate Cancer (mCRPC) and Advanced Salivary Gland Cancers (SGC)
Brief Title: P-PSMA-101 CAR-T Cells in the Treatment of Subjects With Metastatic Castration-Resistant Prostate Cancer (mCRPC) and Advanced Salivary Gland Cancers (SGC)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study closed
Sponsor: Poseida Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: P-PSMA-101-001
Record Dates: First submitted 2020-01-28; First posted 2020-01-31 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-01

CONDITIONS: Prostatic Neoplasms, Castration-Resistant; Neoplasms by Histologic Type; Neoplasms, Prostate; Prostate Cancer; Metastatic Castration-resistant Prostate Cancer; Neoplasms; Prostatic Neoplasms; Genital Neoplasms, Male; Urogenital Neoplasms; Neoplasms by Site; Prostatic Disease; Salivary Gland Cancer; Salivary Gland Tumor; Adenoid Cystic Carcinoma; Salivary Duct Carcinoma; Mucoepidermoid Carcinoma; Acinic Cell Tumor
Keywords: CAR-T cells; metastatic castration-resistant prostate cancer (mCRPC)
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant; Neoplasms by Histologic Type; Prostatic Neoplasms; Neoplasms; Genital Neoplasms, Male; Urogenital Neoplasms; Neoplasms by Site; Prostatic Diseases; Salivary Gland Neoplasms; Carcinoma, Adenoid Cystic; Carcinoma, Mucoepidermoid; Carcinoma, Acinar Cell

STUDY DESIGN:
Intervention Model Description: Open label, 3 + 3 design of dose-escalating cohorts with open label, dose expansion at RP2D
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- P-PSMA-101 CAR-T cells (Single Dose - Part 1a) (Experimental): Single ascending dose cohorts, given in a single intravenous infusion of CAR-T cells, following conditioning chemotherapy regimen A. Rimiducid may be administered as indicated.
  Interventions: Biological: P-PSMA-101 CAR-T cells; Drug: Rimiducid
- P-PSMA-101 CAR-T cells (Multiple Dose - Part 1b) (Experimental): Cyclic administration of ascending dose cohorts, given in a single intravenous infusion of CAR-T cells, following conditioning chemotherapy regimen A. Rimiducid may be administered as indicated.
  Interventions: Biological: P-PSMA-101 CAR-T cells; Drug: Rimiducid
- P-PSMA-101 CAR-T cells (Single Dose - Part 1c) (Experimental): Single ascending dose cohorts, given in a single intravenous infusion of CAR-T cells, following conditioning chemotherapy regimen B. Rimiducid may be administered as indicated.
  Interventions: Biological: P-PSMA-101 CAR-T cells; Drug: Rimiducid
- P-PSMA-101 CAR-T cells (Multiple Dose - Part 1d) (Experimental): Cyclic administration of ascending dose cohorts, given via intravenous infusions of CAR-T cells, following conditioning chemotherapy regimen B. Rimiducid may be administered as indicated.
  Interventions: Biological: P-PSMA-101 CAR-T cells; Drug: Rimiducid

INTERVENTIONS:
Biological: P-PSMA-101 CAR-T cells — P-PSMA-101 is an autologous chimeric antigen receptor (CAR) T-cell therapy designed to target prostate cancer cells expressing the cell surface antigen prostate-specific membrane antigen (PSMA).
Drug: Rimiducid — Rimiducid (safety switch activator) may be administered as indicated

SUMMARY:
An open-label, multi-center, single and cyclic ascending dose study of P-PSMA-101 autologous CAR-T cells in patients with mCRPC and SGC.

DETAILED DESCRIPTION:
This is an open label, multi-center Phase 1 study that will follow a 3 + 3 design of dose-escalating cohorts of single and multiple doses of P-PSMA-101 to determine a Recommended Phase 2 Dose (RP2D). Additional participants will be treated with P-PSMA-101 at the determined RP2D.

Following consent, enrolled participants will undergo a leukapheresis procedure to obtain peripheral blood mononuclear cells (PBMCs) which will be sent to a manufacturing site to produce P-PSMA-101 CAR-T cells. The cells will then be returned to the investigational site and administered after a lymphodepleting chemotherapy regimen. Rimiducid may be administered as indicated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥18 years of age
* Must have a confirmed diagnosis of mCRPC or SGC
* Must have measurable disease by RECIST 1.1 or bone only metastases with measurable PSA (≥1 ng/mL) (mCRPC subjects only)
* Must have progressed by PCWG3 and/or RECIST 1.1 (mCRPC subjects only)
* Must be willing to practice birth control from screening and for 2 years after the last administration of P-PSMA-101
* Must have adequate vital organ function within pre-determined parameters
* Must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1

Exclusion Criteria:

* Has inadequate venous access and/or contraindications to leukapheresis
* Has an active second malignancy in addition to mCRPC or SGC, excluding low-risk neoplasms such as non-metastatic basal cell or squamous cell skin carcinoma
* Has a history of or active autoimmune disease
* Has a history of significant central nervous system (CNS) disease, such as stroke or epilepsy
* Has an active systemic (viral, bacterial or fungal) infection
* Has received anti-cancer medications (excluding GnRH targeted therapies) within 2 weeks of the time of initiating conditioning chemotherapy
* Has received immunosuppressive medications (including anti-cancer medications) within 2 weeks of initiating leukapheresis and/or expected to require them while enrolled in the study
* Has received systemic corticosteroid therapy within 2 weeks of either the required leukapheresis or is expected to require it during the course of the study
* Has CNS metastases or symptomatic CNS involvement
* Has a history of significant ocular disease
* Has a history of significant liver disease or active liver disease
* Has liver metastases (<5 lesions and maximum diameter </= 2.5 cm permitted)
* Has a history of or known predisposition to HLH or MAS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Assess the Safety of P-PSMA-101 | Baseline through 15 years
  Incidence and severity of treatment-emergent adverse events
Determine the maximum tolerated dose of P-PSMA-101 | Baseline through Day 28
  Rate of dose limiting toxicities (DLT)
Assess the efficacy of P-PSMA-101 (ORR) | Baseline through 15 years
  According to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, secondarily Immune Response Evaluation Criteria in Solid Tumors (iRECIST), and Prostate Cancer Response assessed by Prostate Cancer Working Group 3 (PCWG3) criteria: Overall Response Rate (ORR)-Percentage of patients with complete response (CR) or partial response (PR).

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Belani, M.D., Study Director — Sponsor Executive Medical Director
Locations (10):
- United States (10):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of California San Diego, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Tulane University Hospital and Clinic, New Orleans, Louisiana
  - University of Maryland, Baltimore, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Tennessee Oncology, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No